CLINICAL TRIAL: NCT05948787
Title: A Multi-site Randomized Controlled Trial: Testing the Feasibility and Effectiveness of the Strong Families Programme in the Philippines, Skills-based Prevention Intervention for Families With Children Ages 8-14 Years Old.
Brief Title: Assessing the Feasibility of Providing a Family Skills Intervention "Strong Families" for Families in the Philippines.
Acronym: SF_RCT_POPHL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: United Nations Office on Drugs and Crime (UNODC) (Other Government)
Collaborators: Polytechnique University of the Philippines (Unknown); Anti-Drug Abuse Councils, LGUs in the Philippines (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: UNODC POPHL 2023; INL US State Department (Other Grant/Funding Number: INL, US State Department)
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-06

CONDITIONS: Parenting Skills; Family Relationship
Keywords: communication; bonding
MeSH Terms: conditions — Communication | interventions — Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: Method
  * Caregivers will complete a battery of questionnaires, right before intervention(Time 1), two weeks post intervention (Time 2) and also six weeks post intervention (Time 3)
  * Semi-Structured interviews with a selected group of parents that have completed the Strong Families programme and facilitators
  Caregiver measures
  1. Family Demographics Questionnaire: FDQ
  2. Strengths and Difficulties Questionnaire: SDQ (Goodman, 1997) - behavioral screening questionnaire (25 items)
  3. Parental and Family Adjustment Scale: PAFAS (Sanders, Morawska, Haslam, Filus & Fletcher, 2014) measures parenting practices and parental adjustment (30 items), this has been developed to be used in low resource settings
  4. (Person Most Knowledgeable) Child and Youth Resilience Measure: PMK-CYRM-R (Jefferies, P., McGarrigle, L., & Ungar, M. (2018)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): Intervention group' Families take part in weekly sessions of Strong Families for 3 weeks. All family's complete measures again (Time 2, two weeks post intervention). All family's complete measures again (Time 3, 6 weeks post intervention)
  Interventions: Behavioral: Psychosocial intervention
- Waitlist group' Families take part in weekly sessions of Strong Families after the data measures (Experimental): Families in the RCT will be randomized to implementation of the Intervention or Waitlist group . Families will be allocated using online software (www.sealedenvelope.com). We are aware that randomization before recruiting participants can influence recruitment and dropout in the control arm. To minimize these issues, we have included costs for compensating families for participation in study measure completion and will instruct staff not to reveal family allocation until families have agreed to take part and before signing informed consent. This is an un-blinded trial. Research assistants, staff and families will be aware of participants' allocated condition during the trial.
  Interventions: Behavioral: Psychosocial intervention

INTERVENTIONS:
Behavioral: Psychosocial intervention — A structured sessions for families that promotes improving communication, bonding, and improved parenting techniques in managing stress within the family setting.
  Other Names: Group sessions

SUMMARY:
The Strong Families Programme was introduced by UNODC in the Philippines in 2018 through the training of facilitators. Twenty-six participants trained in the program from different cities and municipalities. Afterward, Caloocan, Marikina, Palawan, Pasig, and Quezon City Local Government Units (LGUs) started to train more facilitators to allow them to pilot the program in their communities. Eventually, these cities and municipalities managed to engage families to benefit from the Strong Families Programme.

The current study aims to explore the feasibility, effectiveness and acceptability of this universal prevention program with families in the Philippines, and the feasibility of delivering the program.

The primary objective will be to test the effectiveness of the Strong Families program in improving family skills outcomes and caregiver and child mental health, as reported by caregivers, when implemented in the Philippines.

The secondary objective will be to calculate the extent of family's attendance of Strong Families sessions, to evaluate completeness of program delivery.

The tertiary objective will be to explore the cultural and contextual acceptability of the Strong Families program for families in the Philippines.

A two-arm feasibility Randomized Controlled Trial with two arms: 1) Implementation of Strong Families (Intervention Group) and 2) Wait list/Control (Services-as-usual). This trial will have an embedded process evaluation.

This study will take place in five locations in the Philippines. The implementation usually happens at the Barangay Level (The smallest administrative division in the Philippines and is the native Filipino term for a village, district, or ward)

DETAILED DESCRIPTION:
Participants will be parents or caregivers and one child and up to two children under their care aged between 8-14 years. recruitment of the families will be done by the LGUs considering the opportunistic, 'universal' approach.

The study will be coordinated with the Anti-drug Abuse Councils at the Local Government Units (LGUs) of the five project sites supported by UNODC that mitigates the negative impact of COVID-19 on at-risk communities in the country. They will communicate the study with the Barangay Captains (Chief of the town) to advertise the study to their respective Barangays. Whether the study is announced via an online platform or through a traditional announcement (roving vehicle with a megaphone), or announcement posters, this will be arranged with the Barangay Captains.

Exclusion criteria

* Families that have taken part in family skills training in the past 24 months
* Families in which parent/caregiver live separately from children
* Families in which parents/caregivers/children identified to have drug dependence

Intervention

Strong Families will be delivered to families in groups of approximately 8 to 12 families. Only one or two parents or main caregivers will be invited to attend with a maximum of two children under their care aged 8-14.

The program consists of three meetings (Table 2), one parent (caregiver pre session, 1 hour) during week one. In week two and three, meetings will be one session in which parents and children will meet individually with facilitators for a parent/child session (1 hour each), then come together at the end for a joint family activity session (1 hour session). The first session (parent pre-session) explores parents' challenges and develops ways to better deal with stress. In week two, parents are taught the value of using both love and limits and listening to children while children are taught how to deal with stress. During the family session they practice positive communication and are encouraged to exercise stress relief techniques together. In week 3, parents are trained on how to encourage good behavior and discourage misbehavior, while children explore rules and responsibilities and think about future goals in addition to the important roles their caregivers play in their lives. In the final family session, caregivers and children come together to learn about family values and are encouraged to share appreciation for each other.

Families in the RCT will be randomized to implementation of the Intervention or Waitlist group. Families will be allocated using online software (www.sealedenvelope.com). We are aware that randomization before recruiting participants can influence recruitment and dropout in the control arm. To minimize these issues, we have included costs for compensating families for participation in study measure completion and will instruct staff not to reveal family allocation until families have agreed to take part and before signing informed consent. This is an un-blinded trial. Research assistants, staff and families will be aware of participants' allocated condition during the trial.

Participant activities within the RCT component of the trial

* Participants who show interest in taking part or are invited by the research team along with their participating child, will be given both written and verbal information about the program participation activities and the evaluation process.
* Those interested will be invited to attend a meeting in which they will complete questionnaires, assisted by a research assistant. This will be the first 'measure completion session' of three. During this meeting, they will sign a consent form.
* Participants will be randomly allocated to the intervention or waitlist/control group
* Families in the intervention group will begin the Strong Families program. (Table 2).
* One week and six weeks after the last session that the Intervention group attended the Strong Families Program, all families (also those from the waitlist group in the RCT) will be invited to a session to complete the same questionnaires they completed at the first 'measure completion session'.
* Participants in the intervention group will be asked if they would like to take part in interviews at the time 2 data collection, as indicated in the timeline in Table 3, and given both written and verbal information about the interview process, including questions to be asked and length of interview. Those that are interested will be enlisted and given the schedule and location of the interview.

ELIGIBILITY:
Inclusion Criteria:

* Parent or caregivers that speak Filipino (Tagalog) with at least one child and up to two children under their care aged 8-14
* Willing to take part in the program
* Will be in town for the duration of the programme and research sessions

Exclusion Criteria:

* Families that have taken part in family skills training in the past 24 months
* Families in which parent/caregiver live separately from children
* Families in which parents/caregivers/children identified to have drug dependence

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Improved parenting skills | three data time frames: 2 weeks post intervention, 3 weeks post intervention, and 6 weeks post intervention
  Improved caregiver confidence in family management skills Improved caregiving in parenting skills Improved child behaviour Reduced aggressive and hostile behaviours Increased capacity to cope with stress Improved mental health outcomes in children and parents

CONTACTS AND LOCATIONS:
Overall Officials: Aala El Khani, Principal Investigator — United Nations Office on Drugs and Crime (UNODC); Wadih Maalouf, Study Director — United Nations Office on Drugs and Crime (UNODC); Olivier Lermet, Study Director — United Nations Office on Drugs and Crime (UNODC); Aimee Rose Manda, PhD, Principal Investigator — Polytechnique University of the Philippines; Geraldine F Santos, PhD, Principal Investigator — Polytechnique University of the Philippines
Locations (5):
- Philippines (5):
  - Caloocan Anti-drug Abuse Council, Caloocan
  - Ministry of Social Services Department, Cotabato City
  - Marikina Anti-drug Abuse Council, Marikina City
  - Anti-drug Abuse Council Office of Pasig, Pasig
  - Quezon City Anti-drug Abuse Council, Quezon City

IPD SHARING:
Plan to Share IPD: No
The project coordinator in the Philippines, Ms. Shella Ruiz-Marquez is responsible for storage of all digital and non-digital data. Interviews will be audio recorded (with participants' and facilitators permission) using a digital voice recorder supporting file encryption. Notes will be written up as soon as possible following observation sessions and stored with transcriptions of digital recordings using (Google Cloud) software. Identifying material will be removed as soon as possible from transcripts and notes. Qualitative data will be copied into software files. Electronic copies of transcripts will be held separately from digital recordings of interviews and the file containing participants' names and corresponding numbers. At the end of the project, all non-digital data will be stored at the UNODC Philippines office for a minimum of 5 years after completion of the study. All digital data will be entered electronically using Epidata software and analysed using commercial statistica

REFERENCES:
- [Background] 1 Prevention, Treatment and Rehabilitation Section, Drug Prevention and Health Branch, United Nations Office on Drugs and Crime (UNODC), Division of Operations, Wagramer Strasse 5, A-1400 Vienna, Austria; karin.haar@un.org (K.H.); wadih.maalouf@un.org (W.M.) 2 Division of Psychology & Mental Health, University of Manchester, Manchester M13 9WL, UK; rachel.calam@manchester.ac.uk * Correspondence: aala.el-khani@un.org
- [Background] Prevention, Treatment and Rehabilitation Section, Drug Prevention and Health Branch, Division of Operations, United Nations Office on Drugs and Crime (UNODC), Wagramer Strasse 5, A-1400 Vienna, Austria; ali.yassine@un.org (A.Y.); karin.haar@un.org (K.H.); wadih.maalouf@un.org (W.M.) 2 Drug Demand Reduction Division, United Nations Office on Drugs and Crime (UNODC), Menara Thamrin Building 10th Floor, Central Jakarta, Jakarta 10250, Indonesia; narendra.narotama@un.org (N.N.); lucky.pramitasari@un.org (L.P.) 3 Charitas Hospital Palembang, Central Jakarta, Jakarta 30129, Indonesia; melvi.rosilawati@gmail.com * Correspondence: aala.el-khani@un.org
- [Background] Prevention, Treatment and Rehabilitation Section, Drug Prevention and Health Branch, Division of Operations, United Nations Office on Drugs and Crime (UNODC), Wagramer Strasse 5, A-1400 Vienna, Austria; Aala.elkhani@gmail.com (A.E.-K.); Karin.haar@un.org (K.H.) 2 United Nations Office on Drugs and Crime, Program Office Serbia, Bulevar Zorana Djindjica 64, 11000 Belgrade, Serbia; Milos.stojanovic@un.org * Correspondence: Wadih.maalouf@un.org † Authors' information: The views expressed in this Article do not necessarily reflect the views of the United Nations or its officials or Member States.
- [Background] Haar K, El-Khani A, Molgaard V, Maalouf W; Afghanistan field implementation team. Strong families: a new family skills training programme for challenged and humanitarian settings: a single-arm intervention tested in Afghanistan. BMC Public Health. 2020 May 7;20(1):634. doi: 10.1186/s12889-020-08701-w. PMID 32381064
- See also: To support breaking the vicious cycle of families reproducing negative coping patterns, the United Nations Office on Drugs and Crime (UNODC) has been implementing a global initiative on prevention piloting evidence-based family skills prevention in low- — https://www.unodc.org/unodc/site-search.html?q=Strong+Families+Programme